CLINICAL TRIAL: NCT05066828
Title: Patient Satisfaction of Conventional One-piece Versus Two-piece Magnet-retained Obturators for Patients With Complete Edentulism: A Crossover Study
Brief Title: Conventional One-piece Versus Two-piece Magnet-retained Obturators
Acronym: obturators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sharaf Mohamed Yahia, lecturer, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 214/2018
Record Dates: First submitted 2021-07-05; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional obturator (Active Comparator): Participants received conventional obturator one piece
  Interventions: Other: two pieces obturator
- sectional obturator (Experimental): two pieces obturators connected by magnet attachments
  Interventions: Other: two pieces obturator

INTERVENTIONS:
Other: two pieces obturator — patient received two pieces obturator connecting by magnet attachment
  Other Names: sectional obturator

SUMMARY:
Evaluation of patients' satisfaction with conventional one-piece obturators versus two pieces magnet -retained obturators in completely edentulous patient maxillectomy cases.

DETAILED DESCRIPTION:
Ten completely edentulous participants with hemimaxillectomy (8 males and 2 females) were selected in an across over study. Participants received conventional obturator one piece and two pieces obturator connecting by magnet attachment in alternate periods (sequences A-B and B-A), and outcomes were assessed after 1 week,3 months, and 6 months Evaluation included Obturator Functioning Scale(OFS) and Oral Health Impact Profile for edentulous people (OHIP-EDENT ). One way ANOVA test and Multivariate analysis of variance with a general linear model with repeated measure was used to test the impact of the group, time, and order on each of the studied scores (α=.05).

ELIGIBILITY:
Inclusion Criteria:

- completely edentulous participants with hemimaxillectomy mouth opening is not less than 25 mm and intact soft palate

Exclusion Criteria:

* exposed to radiotherpy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | 1 week to 6 months
  evaluation of satisfaction by Obturator Functioning Scale(OFS)

SECONDARY OUTCOMES:
patient satisfaction | 1 week to 6 months
  evaluation of satisfaction by Oral Health Impact Profile for edentulous people (OHIP-EDENT )

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided